CLINICAL TRIAL: NCT01436682
Title: Assisted Nerve Blocks
Status: Completed | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Thomas Hemmerling, Associate Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: GEN11-073
Record Dates: First submitted 2011-09-19; First posted 2011-09-20 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Surgery
Keywords: Nerve Blocks

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study investigates assisted nerve blocks using an ultrasound machine.

ELIGIBILITY:
Inclusion Criteria:

* indication for nerve blocks

Exclusion Criteria:

* patient not able to provide the informed consent
* allergy to local anesthetics

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient undergoing surgery which necessitates a peripheral nerve block to relieve postoperative pain.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2011-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Feasability of assisted nerve blocks | 24h

CONTACTS AND LOCATIONS:
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada